CLINICAL TRIAL: NCT07233070
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Safety and Efficacy of HRS-7450 Injection in Patients With Acute Ischemic Stroke.
Brief Title: HRS-7450 Injection Phase II Clinical Trial for Acute Ischemic Stroke.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-7450-201
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A: HRS-7450 Injection (Experimental)
  Interventions: Drug: HRS-7450 Injection
- Treatment group B: HRS-7450 Injection (Experimental)
  Interventions: Drug: HRS-7450 Injection
- Treatment group C: HRS-7450 Injection (Experimental)
  Interventions: Drug: HRS-7450 Injection
- Treatment group D: HRS-7450 Injection Placebo. (Placebo Comparator)
  Interventions: Drug: HRS-7450 Injection Placebo

INTERVENTIONS:
Drug: HRS-7450 Injection — HRS-7450 Injection; low dose
  Arms: Treatment group A: HRS-7450 Injection
Drug: HRS-7450 Injection — HRS-7450 Injection; Intermediate dose
  Arms: Treatment group B: HRS-7450 Injection
Drug: HRS-7450 Injection — HRS-7450 Injection; high dose
  Arms: Treatment group C: HRS-7450 Injection
Drug: HRS-7450 Injection Placebo — HRS-7450 Injection Placebo
  Arms: Treatment group D: HRS-7450 Injection Placebo.

SUMMARY:
This study plans to enroll a total of 208 patients with Acute Ischemic Stroke (AIS) who present within 4.5 to 24 hours of symptom onset and meet the specified imaging criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand and voluntarily participate in this study, and sign the informed consent form;
2. Aged between 18 and 80 years inclusive (18 ≤ age ≤ 80), regardless of gender;
3. Onset of symptoms within 4.5 to 24 hours;
4. Clinically diagnosed with acute ischemic stroke;
5. Pre-stroke modified Rankin Scale (mRS) score < 2;
6. National Institutes of Health Stroke Scale (NIHSS) score between 6 and 25 (inclusive) at screening;
7. Meet the imaging inclusion criteria;
8. Female subjects of childbearing potential and male subjects with partners of childbearing potential must use highly effective contraception and avoid sperm/ova donation.

Exclusion Criteria:

1. Treatment with thrombolytic therapy.
2. Planned endovascular therapy.
3. Arterial dissection of the head, neck, or aorta.
4. Multiple infarctions across multiple large vascular territories.
5. NIHSS level of consciousness item 1a score > 2.
6. Neurological deficits presenting after a seizure or post-ictal state, or the presence of other neurological conditions leading to uncooperative or unwillingness to cooperate with examination.
7. Hypodensity exceeding one-third of the middle cerebral artery (MCA) territory on non-contrast CT scan.
8. Intracranial tumor, arteriovenous malformation (AVM), or giant aneurysm.
9. History of intracranial hemorrhagic disease, including but not limited to intracerebral hemorrhage, subarachnoid hemorrhage, etc.
10. History of ischemic stroke, severe head trauma, or intracranial/intraspinal surgery within the past 3 months.
11. Visceral bleeding within the past 3 weeks, including but not limited to gastrointestinal or genitourinary bleeding.
12. Major surgery or severe trauma within the past 2 weeks.
13. Arterial puncture at a non-compressible site within the past week.
14. Systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥100 mmHg despite aggressive antihypertensive treatment.
15. Known significant bleeding tendency or severe coagulation disorder.
16. Blood glucose at screening >22.2 mmol/L or <2.8 mmol/L; subjects may be re-evaluated after active treatment.
17. Within the past 3 months: acute ST-segment elevation myocardial infarction (MI), and/or acute decompensated heart failure, and/or QTc > 520 ms, and/or hospitalization for acute coronary syndrome, MI, cardiac arrest, or unplanned coronary intervention; or New York Heart Association (NYHA) Class III/IV heart failure; or known ventricular tachycardia.
18. Significant liver disease history, or AST and/or ALT and/or GGT ≥3 × ULN, and/or total bilirubin (TBIL) ≥2 × ULN, or known congenital disorder of bilirubin metabolism.
19. Clinically significant severe renal disease, or estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m².
20. History of hemolytic anemia due to various causes, currently under treatment or not meeting cure criteria.
21. Known allergy or hypersensitivity to HRS-7450 or any excipients in its formulation.
22. Treatment with therapeutic doses of heparin or low molecular weight heparin within 24 hours.
23. Use of oral anticoagulants within 48 hours, including vitamin K antagonists, direct thrombin inhibitors, factor Xa inhibitors, or other investigational anticoagulants.
24. Use of glycoprotein IIb/IIIa receptor inhibitors within 48 hours.
25. Female subjects who are pregnant or breastfeeding, or with a positive pregnancy test.
26. Participation in another drug or device clinical trial within the 3 months prior to screening.
27. Terminal illness with a life expectancy of less than 1 year.
28. Any other condition deemed by the investigator to make the subject unsuitable for participation in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
mRS score of 0-1 at 90 days | within 90 days after the start of administration

SECONDARY OUTCOMES:
Reperfusion rate at 24 hours; | within 24 hours after the start of administration
Recanalization rate at 24 hours; | within 24 hours after the start of administration
Proportion of subjects with ≥8-point reduction in NIHSS score or NIHSS score of 0-1 at 24 hours; | within 24 hours after the start of administration
Infarct volume at 7 days; | within 7 days after the start of administration
Proportion of subjects with ≥8-point reduction in NIHSS score or NIHSS score of 0-1 at 7 days; | within 7 days after the start of administration
NIHSS score at 14 days; | within 14 days after the start of administration
mRS score at 90 days; | within 90 days after the start of administration
Proportion of subjects with mRS score 0-2 at 90 days; | within 90 days after the start of administration
Incidence of symptomatic intracranial hemorrhage (sICH) within 36 hours after dosing; | within 36 hours after the start of administration
Incidence of symptomatic intracranial hemorrhage (sICH) within 7 days after dosing; | within 7 days after the start of administration
Incidence of intracranial hemorrhage (ICH) within 36 hours after dosing; | within 36 hours after the start of administration
Incidence of intracranial hemorrhage (ICH) within 7 days after dosing; | within 7 days after the start of administration
Incidence of major non-intracranial hemorrhage within 36 hours after dosing; | within 36 hours after the start of administration
Incidence of major non-intracranial hemorrhage within 7 days after dosing; | within 7 days after the start of administration
Mortality rate at 7 days after dosing; | within 7 days after the start of administration
Mortality rate at 90 days after dosing; | within 90 days after the start of administration

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Linyi People's Hospital, Linyi, Shandong

IPD SHARING:
Plan to Share IPD: Undecided